CLINICAL TRIAL: NCT06261333
Title: Influence of Telangiectasia and Anemia on the Well-being and Quality of Life of Patients With Hereditary Hemorrhagic Telangiectasia (HHT).
Brief Title: Quality of Life in Patients With Hemorrhagic Telangiectasia
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Essen (Other)
Responsible Party: Principal Investigator, Freya Droege, Principal Investigator, University Hospital, Essen
Other Study IDs: 23-11519-BO
Record Dates: First submitted 2024-01-12; First posted 2024-02-15 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Hereditary Hemorrhagic Telangiectasia
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaires — No Intervention

SUMMARY:
Hereditary Hemorrhagic Telangiectasia (HHT), also known as Osler's disease, is a genetic disorder that leads to abnormal blood vessel formations. It primarily affects blood vessels in the skin, mucous membranes, and internal organs. The disease can be clinically diagnosed using the Curaçao criteria (1. Positive family history of HHT, 2. Recurrent and spontaneous epistaxis, 3. Multiple typical telangiectasias, 4. Organ involvement with vascular malformations, especially in the liver, lungs, gastrointestinal tract, or brain); if a patient meets at least 3 criteria, the diagnosis of HHT can be established.

Patients with HHT often have telangiectasias on their faces. Additionally, many patients suffer from anemia, which can result in a pale and potentially tired appearance. Patients with HHT may be less satisfied with their appearance due to the aesthetic changes in their faces and may also experience psychosocial impairment. To further investigate this, various validated questionnaires (FACE-Q©, PROMIS-Profile-29+2, EQ5D), as well as routinely collected clinical data (e.g., laboratory values including hemoglobin levels, Curaçao criteria, smoking status, alcohol consumption, and the Epistaxis Severity Score (ESS)) will be used.

ELIGIBILITY:
Inclusion criteria:

* knowledge of german language
* Age above 17 years
* capable of giving consent
* Diagnosis of HHT (Curaçao criteria or genetic testing)

Exclusion criteria:

-Individuals not meeting the inclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from HHT
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of Life and Patient Satisfaction measured using the FACE-Questionnaire | one year
  Using patient reported outcome measurements: Face-Questionnaire and Patient-Reported Outcomes Measurement Information System (PROMIS) in order to assess the quality of life in patients with HHT

CONTACTS AND LOCATIONS:
Locations (1):
- Departement of Otorhinolaryngology - Head and Neck Surgery University Hospital Essen, Essen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analysed during the current study are available on reasonable request